CLINICAL TRIAL: NCT02465567
Title: A Randomized, Double-Blind, Multi-Center, Parallel-Group Study to Assess the Efficacy and Safety of PT010 Relative to PT003 and PT009 on COPD Exacerbations Over a 52-Week Treatment Period in Subjects With Moderate to Very Severe COPD (Ethos)
Brief Title: Study to Assess the Efficacy and Safety of PT010 Relative to PT003 and PT009 in Subjects With Moderate to Very Severe COPD (Ethos)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pearl Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PT010005
Record Dates: First submitted 2015-05-29; First posted 2015-06-08 (Estimated); Results first posted 2021-02-02 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2021-01

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- BGF (PT010) MDI 320/14.4/9.6 μg (Experimental): BGF MDI 320/14.4/9.6 μg, Budesonide, Glycopyrronium, Formoterol Fumarate Aerosol (PT010, BGF metered dose inhaler [MDI])
  Interventions: Drug: BGF MDI 320/14.4/9.6 μg
- BGF (PT010) MDI 160/14.4/9.6 μg (Experimental): BGF MDI 160/14.4/9.6 μg, Budesonide, Glycopyrronium, Formoterol Fumarate Aerosol (PT010, BGF metered dose inhaler [MDI])
  Interventions: Drug: BGF MDI 160/14.4/9.6 μg
- BFF (PT009) MDI 320/9.6 μg (Experimental): BFF MDI 320/9.6 μg Budesonide, Formoterol Fumarate Aerosol Glycopyrronium and Formoterol Fumarate Inhalation Aerosol (PT009)
  Interventions: Drug: BFF MDI 320/9.6 μg
- GFF (PT003) MDI 14.4/9.6 μg (Experimental): GFF MDI 14.4/9.6 μg Glycopyrronium, Formoterol Fumarate Aerosol Budesonide and Formoterol Fumarate Inhalation Aerosol (PT003)
  Interventions: Drug: GFF MDI 14.4/9.6 μg

INTERVENTIONS:
Drug: BGF MDI 320/14.4/9.6 μg — Budensonide, Glycopyrronium, and Formoterol Fumarate
  Other Names: BGF
  Arms: BGF (PT010) MDI 320/14.4/9.6 μg
Drug: GFF MDI 14.4/9.6 μg — Glycopyrronium, and Formoterol Fumarate
  Other Names: GFF
  Arms: GFF (PT003) MDI 14.4/9.6 μg
Drug: BGF MDI 160/14.4/9.6 μg — Budensonide, Glycopyrronium, and Formoterol Fumarate
  Other Names: BGF
  Arms: BGF (PT010) MDI 160/14.4/9.6 μg
Drug: BFF MDI 320/9.6 μg — Budensonide, and Formoterol Fumarate
  Other Names: BFF
  Arms: BFF (PT009) MDI 320/9.6 μg

SUMMARY:
This is a randomized, double-blind, multi-center, parallel-group study to assess the efficacy and safety of PT010 relative to PT003 and PT009 on COPD exacerbations subjects with moderate to very severe COPD.

DETAILED DESCRIPTION:
A randomized, double-blind, multi-center, parallel-group study to assess the efficacy and safety of PT010 relative to PT003 and PT009 on COPD exacerbations over a 52-week treatment period in subjects with moderate to very severe COPD.

ELIGIBILITY:
Inclusion Criteria

* Non-child bearing potential (ie, physiologically incapable of becoming pregnant, including any female who is 2 years post-menopausal); or Child bearing potential, has a negative serum pregnancy test at Visit 1, and agrees to acceptable contraceptive methods used consistently and correctly for the duration of the study.
* Subjects with an established clinical history of COPD as defined by the American Thoracic Society (ATS)/European Respiratory Society (ERS),
* Current or former smokers with a history of at least 10 pack-years of cigarette smoking.
* Forced expiratory volume in 1 second (FEV1)/Forced vital capacity (FVC) ratio must be <0.70 and FEV1 must be <65% predicted normal value calculated using NHANES III reference equations (or reference norms applicable to other regions).
* Subjects with history of exacerbations.

Please refer to the study protocol for the complete inclusion criteria list.

Exclusion Criteria

* Significant diseases or conditions other than COPD, which, in the opinion of the Investigator, may put the subject at risk because of participation in the study or may influence either the results of the study or the subject's ability to participate in the study.
* Women who are pregnant or lactating, or are planning to become pregnant during the course of the study, or women of childbearing potential who are not using an acceptable method of contraception.
* Subjects, who in the opinion of the Investigator, have a current diagnosis of asthma.
* Subjects who have been hospitalized due to poorly controlled COPD within 3 months prior to Visit 1 (Screening)
* Subjects who have poorly controlled COPD, defined as acute worsening of COPD that requires treatment with oral corticosteroids or antibiotics within 6 weeks prior to Visit 1 (Screening)
* Immune suppression or severe neurological disorders affecting control of the upper airway or other risk factors that in the opinion of the Investigator would put the subject at substantial risk of pneumonia.
* Subjects with a diagnosis of narrow angle glaucoma, who, in the opinion of the Investigator, have not been adequately treated.
* Subjects who have a history of hypersensitivity to β2-agonists, budesonide or any other corticosteroid components, glycopyrronium or other muscarinic anticholinergics, or any other component of the IMPs.

Please refer to the study protocol for the complete inclusion criteria list.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8588 (Actual)
Dates: Start 2015-06-30 (Actual); Primary Completion 2019-07-26 (Actual); Study Completion 2019-07-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul M Dorinsky, MD, Study Director — Pearl Therapeutics
Locations (566):
- United States (252):
  - Research Site, Andalusia, Alabama
  - Research Site, Athens, Alabama
  - Research Site, Birmingham, Alabama
  - Research Site, Dothan, Alabama
  - Research Site, Florence, Alabama
  - Research Site, Foley, Alabama
  - Research Site, Gulf Shores, Alabama
  - Research Site, Jasper, Alabama
  - Research Site, Mobile, Alabama
  - Research Site, Montgomery, Alabama
  - Research Site, Scottsboro, Alabama
  - Research Site, Sheffield, Alabama
  - Research Site, Peoria, Arizona
  - Research Site, Phoenix, Arizona
  - Research Site, Scottsdale, Arizona
  - Research Site, Conway, Arkansas
  - Research Site, Little Rock, Arkansas
  - Research Site, North Little Rock, Arkansas
  - Research Site, Bakersfield, California
  - Research Site, Beverly Hills, California
  - Research Site, Cerritos, California
  - Research Site, El Cajon, California
  - Research Site, Escondido, California
  - Research Site, Fresno, California
  - Research Site, Gold River, California
  - Research Site, Hawaiian Gardens, California
  - Research Site, Huntington Beach, California
  - Research Site, Huntington Park, California
  - Research Site, La Mirada, California
  - Research Site, Lakewood, California
  - Research Site, Los Angeles, California
  - Research Site, Newport Beach, California
  - Research Site, Northridge, California
  - Research Site, Palm Springs, California
  - Research Site, Poway, California
  - Research Site, Quartz Hill, California
  - Research Site, Rancho Mirage, California
  - Research Site, Riverside, California
  - Research Site, Rolling Hills Estates, California
  - Research Site, Sacramento, California
  - Research Site, San Diego, California
  - Research Site, Santa Ana, California
  - Research Site, Santa Monica, California
  - Research Site, Stockton, California
  - Research Site, Torrance, California
  - Research Site, Tustin, California
  - Research Site, Upland, California
  - Research Site, Westminster, California
  - Research Site, Wildomar, California
  - Research Site, Colorado Springs, Colorado
  - Research Site, Fort Collins, Colorado
  - Research Site, Lafayette, Colorado
  - Research Site, Boynton Beach, Florida
  - Research Site, Brandon, Florida
  - Research Site, Clearwater, Florida
  - Research Site, Clermont, Florida
  - Research Site, Coral Gables, Florida
  - Research Site, Daytona Beach, Florida
  - Research Site, Fort Lauderdale, Florida
  - Research Site, Gainesville, Florida
  - Research Site, Hialeah, Florida
  - Research Site, Hollywood, Florida
  - Research Site, Homestead, Florida
  - Research Site, Kissimmee, Florida
  - Research Site, Leesburg, Florida
  - Research Site, Loxahatchee Groves, Florida
  - Research Site, Miami, Florida
  - Research Site, Miami Lakes, Florida
  - Research Site, Ormond Beach, Florida
  - Research Site, Panama City, Florida
  - Research Site, Pembroke Pines, Florida
  - Research Site, Pensacola, Florida
  - Research Site, Port Charlotte, Florida
  - Research Site, Sarasota, Florida
  - Research Site, St. Petersburg, Florida
  - Research Site, Tampa, Florida
  - Research Site, Winter Park, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Blue Ridge, Georgia
  - Research Site, Columbus, Georgia
  - Research Site, Dacula, Georgia
  - Research Site, Duluth, Georgia
  - Research Site, Lawrenceville, Georgia
  - Research Site, Norcross, Georgia
  - Research Site, Rincon, Georgia
  - Research Site, Riverdale, Georgia
  - Research Site, Savannah, Georgia
  - Research Site, Woodstock, Georgia
  - Research Site, Belleville, Illinois
  - Research Site, Champaign, Illinois
  - Research Site, Chicago, Illinois
  - Research Site, O'Fallon, Illinois
  - Research Site, Skokie, Illinois
  - Research Site, Michigan City, Indiana
  - Research Site, Valparaiso, Indiana
  - Research Site, Council Bluffs, Iowa
  - Research Site, West Des Moines, Iowa
  - Research Site, Fort Mitchell, Kentucky
  - Research Site, Owensboro, Kentucky
  - Research Site, Paducah, Kentucky
  - Research Site, Crowley, Louisiana
  - Research Site, Lafayette, Louisiana
  - Research Site, Lake Charles, Louisiana
  - Research Site, New Orleans, Louisiana
  - Research Site, Opelousas, Louisiana
  - Research Site, Sunset, Louisiana
  - Research Site, Zachary, Louisiana
  - Research Site, Bangor, Maine
  - Research Site, Baltimore, Maryland
  - Research Site, Columbia, Maryland
  - Research Site, White Marsh, Maryland
  - Research Site, Marlborough, Massachusetts
  - Research Site, Methuen, Massachusetts
  - Research Site, North Dartmouth, Massachusetts
  - Research Site, Buckley, Michigan
  - Research Site, Cadillac, Michigan
  - Research Site, Canton, Michigan
  - Research Site, Caro, Michigan
  - Research Site, Farmington Hills, Michigan
  - Research Site, Flint, Michigan
  - Research Site, Port Huron, Michigan
  - Research Site, Rochester, Michigan
  - Research Site, Southfield, Michigan
  - Research Site, Troy, Michigan
  - Research Site, Edina, Minnesota
  - Research Site, Fridley, Minnesota
  - Research Site, Minneapolis, Minnesota
  - Research Site, Woodbury, Minnesota
  - Research Site, Biloxi, Mississippi
  - Research Site, Belton, Missouri
  - Research Site, Chesterfield, Missouri
  - Research Site, Saint Charles, Missouri
  - Research Site, St Louis, Missouri
  - Research Site, Billings, Montana
  - Research Site, Bellevue, Nebraska
  - Research Site, Las Vegas, Nevada
  - Research Site, Reno, Nevada
  - Research Site, Portsmouth, New Hampshire
  - Research Site, Marlton, New Jersey
  - Research Site, Toms River, New Jersey
  - Research Site, Bronxville, New York
  - Research Site, Brooklyn, New York
  - Research Site, Jamaica, New York
  - Research Site, New Windsor, New York
  - Research Site, New York, New York
  - Research Site, The Bronx, New York
  - Research Site, Asheville, North Carolina
  - Research Site, Burlington, North Carolina
  - Research Site, Charlotte, North Carolina
  - Research Site, Elizabeth City, North Carolina
  - Research Site, Gastonia, North Carolina
  - Research Site, Greensboro, North Carolina
  - Research Site, Hendersonville, North Carolina
  - Research Site, Hickory, North Carolina
  - Research Site, Huntersville, North Carolina
  - Research Site, Lenoir, North Carolina
  - Research Site, Monroe, North Carolina
  - Research Site, Mooresville, North Carolina
  - Research Site, Morganton, North Carolina
  - Research Site, Mount Airy, North Carolina
  - Research Site, New Bern, North Carolina
  - Research Site, Raleigh, North Carolina
  - Research Site, Shelby, North Carolina
  - Research Site, Whiteville, North Carolina
  - Research Site, Wilmington, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Fargo, North Dakota
  - Research Site, Blue Ash, Ohio
  - Research Site, Cincinnati, Ohio
  - Research Site, Columbus, Ohio
  - Research Site, Dayton, Ohio
  - Research Site, Dublin, Ohio
  - Research Site, Kettering, Ohio
  - Research Site, Maumee, Ohio
  - Research Site, Toledo, Ohio
  - Research Site, Edmond, Oklahoma
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Tulsa, Oklahoma
  - Research Site, Medford, Oregon
  - Research Site, Portland, Oregon
  - Research Site, Altoona, Pennsylvania
  - Research Site, Erie, Pennsylvania
  - Research Site, Monroeville, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Phoenixville, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Scottdale, Pennsylvania
  - Research Site, Uniontown, Pennsylvania
  - Research Site, East Providence, Rhode Island
  - Research Site, Providence, Rhode Island
  - Research Site, Anderson, South Carolina
  - Research Site, Charleston, South Carolina
  - Research Site, Columbia, South Carolina
  - Research Site, Easley, South Carolina
  - Research Site, Gaffney, South Carolina
  - Research Site, Greenville, South Carolina
  - Research Site, Greer, South Carolina
  - Research Site, Hodges, South Carolina
  - Research Site, Lancaster, South Carolina
  - Research Site, Mt. Pleasant, South Carolina
  - Research Site, Old Point Station, South Carolina
  - Research Site, Rock Hill, South Carolina
  - Research Site, Seneca, South Carolina
  - Research Site, Spartanburg, South Carolina
  - Research Site, Union, South Carolina
  - Research Site, Rapid City, South Dakota
  - Research Site, Chattanooga, Tennessee
  - Research Site, Hendersonville, Tennessee
  - Research Site, Johnson City, Tennessee
  - Research Site, Knoxville, Tennessee
  - Research Site, Arlington, Texas
  - Research Site, Boerne, Texas
  - Research Site, Carrollton, Texas
  - Research Site, Corsicana, Texas
  - Research Site, Cypress, Texas
  - Research Site, Duncanville, Texas
  - Research Site, El Paso, Texas
  - Research Site, Fort Worth, Texas
  - Research Site, Houston, Texas
  - Research Site, Huntsville, Texas
  - Research Site, Katy, Texas
  - Research Site, Kerrville, Texas
  - Research Site, Killeen, Texas
  - Research Site, Kingwood, Texas
  - Research Site, Lampasas, Texas
  - Research Site, Lewisville, Texas
  - Research Site, Longview, Texas
  - Research Site, Lufkin, Texas
  - Research Site, McKinney, Texas
  - Research Site, Pearland, Texas
  - Research Site, Pflugerville, Texas
  - Research Site, Plano, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Sealy, Texas
  - Research Site, Sherman, Texas
  - Research Site, Splendora, Texas
  - Research Site, The Woodlands, Texas
  - Research Site, Webster, Texas
  - Research Site, Midvale, Utah
  - Research Site, Salt Lake City, Utah
  - Research Site, Abingdon, Virginia
  - Research Site, Burke, Virginia
  - Research Site, Newport News, Virginia
  - Research Site, Richmond, Virginia
  - Research Site, Virginia Beach, Virginia
  - Research Site, Williamsburg, Virginia
  - Research Site, Bellevue, Washington
  - Research Site, Richland, Washington
  - Research Site, Spokane, Washington
  - Research Site, Tacoma, Washington
  - Research Site, Morgantown, West Virginia
  - Research Site, Greenfield, Wisconsin
- Argentina (23):
  - Research Site, Buenos Aires
  - Research Site, CABA
  - Research Site, Capital Federal
  - Research Site, Ciudad Autonoma de Buenos Aire
  - Research Site, Ciudad Autonomade Buenos Aires
  - Research Site, Ciudad Autónoma de Bs. As.
  - Research Site, Ciudad Capital
  - Research Site, Ciudad de Buenos Aire
  - Research Site, Córdoba
  - Research Site, Florida
  - Research Site, La Plata
  - Research Site, Lanús
  - Research Site, Mar del Plata
  - Research Site, Mendoza
  - Research Site, Monte Grande
  - Research Site, Paraná
  - Research Site, Quilmes
  - Research Site, Rosario
  - Research Site, San Fernando
  - Research Site, San Juan Bautista
  - Research Site, San Miguel de Tucumán
  - Research Site, Santa Fe
  - Research Site, Santa Rosa
- Australia (11):
  - Research Site, Adelaide
  - Research Site, Bedford Park
  - Research Site, Box Hill
  - Research Site, Cairns
  - Research Site, Concord
  - Research Site, Everton Park
  - Research Site, Kent Town
  - Research Site, Murdoch
  - Research Site, Nedlands
  - Research Site, South Brisbane
  - Research Site, Westmead
- Austria (8):
  - Research Site, Feldbach
  - Research Site, Grieskirchen
  - Research Site, Hallein
  - Research Site, Linz
  - Research Site, Salzburg
  - Research Site, Thalheim
  - Research Site, Vienna
  - Research Site, Wels
- Belgium (9):
  - Research Site, Brussels
  - Research Site, Erpent
  - Research Site, Genk
  - Research Site, Gilly
  - Research Site, Halen
  - Research Site, Ham
  - Research Site, Lebbeke
  - Research Site, Montigny-le-Tilleul
  - Research Site, Wetteren
- Canada (22):
  - Research Site, Edmonton, Alberta
  - Research Site, Sherwood Park, Alberta
  - Research Site, Vancouver, British Columbia
  - Research Site, Vancouver, CA
  - Research Site, Winnipeg, Manitoba
  - Research Site, Truro, Nova Scotia
  - Research Site, Ajax, Ontario
  - Research Site, Burlington, Ontario
  - Research Site, Greater Sudbury, Ontario
  - Research Site, Hamilton, Ontario
  - Research Site, Mississauga, Ontario
  - Research Site, Sarnia, Ontario
  - Research Site, Windsor, Ontario
  - Research Site, Gatineau, Quebec
  - Research Site, Lévis, Quebec
  - Research Site, Mirabel, Quebec
  - Research Site, Montreal, Quebec
  - Research Site, Pointe-Claire, Quebec
  - Research Site, Québec, Quebec
  - Research Site, Saint-Charles-Borromée, Quebec
  - Research Site, Saint-Jérôme, Quebec
  - Research Site, Saskatoon, Saskatchewan
- Chile (7):
  - Research Site, Concepción
  - Research Site, Curicó
  - Research Site, Quillota
  - Research Site, Santiago
  - Research Site, Talca
  - Research Site, Valparaíso
  - Research Site, Viña del Mar
- China (24):
  - Research Site, Baotou
  - Research Site, Beijing
  - Research Site, Changsha
  - Research Site, Chengdu
  - Research Site, Guangzhou
  - Research Site, Guiyang
  - Research Site, Haikou
  - Research Site, Hangzhou
  - Research Site, Hohhot
  - Research Site, Lanzhou
  - Research Site, Linhai
  - Research Site, Nanchang
  - Research Site, Nanjing
  - Research Site, Pingxiang
  - Research Site, Shanghai
  - Research Site, Shenyang
  - Research Site, Shenzhen
  - Research Site, Shijiazhuang
  - Research Site, Wuhan
  - Research Site, Xi'an
  - Research Site, Xiangtan
  - Research Site, Xuzhou
  - Research Site, Yanji
  - Research Site, Zhanjiang
- Czechia (9):
  - Research Site, Benešov
  - Research Site, Beroun
  - Research Site, Jindřichův Hradec
  - Research Site, Liberec
  - Research Site, Mělník
  - Research Site, Moravský Krumlov
  - Research Site, Prague
  - Research Site, Teplice
  - Research Site, Žatec
- France (5):
  - Research Site, Lyon
  - Research Site, Marseille
  - Research Site, Nantes
  - Research Site, Nîmes
  - Research Site, Vandœuvre-lès-Nancy
- Germany (49):
  - Research Site, Aschaffenburg
  - Research Site, Augsburg
  - Research Site, Bad Wörishofen
  - Research Site, Bamberg
  - Research Site, Bergisch Gladbach
  - Research Site, Berlin
  - Research Site, Bonn
  - Research Site, Cologne
  - Research Site, Cottbus
  - Research Site, Darmstadt
  - Research Site, Deggendorf
  - Research Site, Deggingen
  - Research Site, Dortmund
  - Research Site, Düren
  - Research Site, Erlangen
  - Research Site, Essen
  - Research Site, Frankfurt
  - Research Site, Frankfurt am Main
  - Research Site, Gelsenkirchen
  - Research Site, Grosshansdof
  - Research Site, Halle
  - Research Site, Hamburg
  - Research Site, Hanover
  - Research Site, Ibbenbueren
  - Research Site, Kiel
  - Research Site, Koblenz
  - Research Site, Landsberg
  - Research Site, Leipzig
  - Research Site, Lübeck
  - Research Site, Magdeburg
  - Research Site, Mainz
  - Research Site, Marburg
  - Research Site, München
  - Research Site, Münster
  - Research Site, Neu-Isenburg
  - Research Site, Peine
  - Research Site, Potsdam
  - Research Site, Radebeul
  - Research Site, Rosenheim
  - Research Site, Rüdersdorf
  - Research Site, Rüsselsheim am Main
  - Research Site, Schleswig
  - Research Site, Schwedt
  - Research Site, Wardenburg
  - Research Site, Weinheim
  - Research Site, Wiesbaden
  - Research Site, Wiesloch
  - Research Site, Witten
  - Research Site, Zerbst
- Hungary (15):
  - Research Site, Balassagyarmat
  - Research Site, Budapest
  - Research Site, Csorna
  - Research Site, Debrecen
  - Research Site, Gödöllő
  - Research Site, Kaposvár
  - Research Site, Kapuvár
  - Research Site, Komárom
  - Research Site, Komló
  - Research Site, Miskolc
  - Research Site, Nyíregyháza
  - Research Site, Siófok
  - Research Site, Százhalombatta
  - Research Site, Szigetszentmiklós
  - Research Site, Törökbálint
- Italy (13):
  - Research Site, Bologna
  - Research Site, Foggia
  - Research Site, Genova
  - Research Site, Messina
  - Research Site, Milan
  - Research Site, Modena
  - Research Site, Napoli
  - Research Site, Palermo
  - Research Site, Parma
  - Research Site, Pisa
  - Research Site, Pordenone
  - Research Site, Roma
  - Research Site, Tradate
- Japan (5):
  - Research Site, Osakasayama-shi
  - Research Site, Sakaide-shi
  - Research Site, Seto-shi
  - Research Site, Shinagawa-ku
  - Research Site, Yanagawa-shi
- Mexico (4):
  - Research Site, Cuautitlán Izcalli
  - Research Site, Guadalajara
  - Research Site, México
  - Research Site, Monterrey
- Netherlands (13):
  - Research Site, Almelo
  - Research Site, Almere Stad
  - Research Site, Beek
  - Research Site, Breda
  - Research Site, Capelle aan den IJssel
  - Research Site, Eindhoven
  - Research Site, Enschede
  - Research Site, Harderwijk
  - Research Site, Heerlen
  - Research Site, Hoorn
  - Research Site, Voerendaal
  - Research Site, Zutphen
  - Research Site, Zwolle
- New Zealand (10):
  - Research Site, Auckland
  - Research Site, Christchurch
  - Research Site, Dunedin
  - Research Site, Greenlane
  - Research Site, Greenlane East
  - Research Site, Hamilton
  - Research Site, Havelock North
  - Research Site, Newtown
  - Research Site, Papatoetoe
  - Research Site, Tauranga
- Peru (5):
  - Research Site, Cusco
  - Research Site, Lima
  - Research Site, Miraflores
  - Research Site, Piura
  - Research Site, Santa Beatriz
- Poland (11):
  - Research Site, Bialystok
  - Research Site, Bydgoszcz
  - Research Site, Poznan
  - Research Site, Ruda Śląska
  - Research Site, Rzeszów
  - Research Site, Skarżysko-Kamienna
  - Research Site, Szczecin
  - Research Site, Tarnów
  - Research Site, Warsaw
  - Research Site, Wroclaw
  - Research Site, Zabrze
- Russia (5):
  - Research Site, Arkhangelsk
  - Research Site, Gatchina
  - Research Site, Moscow
  - Research Site, Saint Petersburg
  - Research Site, Yekaterinburg
- Serbia (5):
  - Research Site, Belgrade
  - Research Site, Kamenitz
  - Research Site, Kragujevac
  - Research Site, Niš
  - Research Site, Valjevo
- South Africa (9):
  - Research Site, Benoni
  - Research Site, Bloemfontein
  - Research Site, Boksburg
  - Research Site, Cape Town
  - Research Site, Durban
  - Research Site, Johannesburg
  - Research Site, Port Elizabeth
  - Research Site, Pretoria
  - Research Site, Umhlanga
- Spain (23):
  - Research Site, A Coruña
  - Research Site, Alcobendas
  - Research Site, Alicante
  - Research Site, Alzira
  - Research Site, Badalona(Barcelona)
  - Research Site, Barcelona
  - Research Site, Cartagena
  - Research Site, Girona
  - Research Site, Laredo
  - Research Site, Lleida
  - Research Site, Madrid
  - Research Site, Marbella (Málaga)
  - Research Site, Mataró
  - Research Site, Málaga
  - Research Site, Mérida (Badajoz)
  - Research Site, Pamplona
  - Research Site, Peralada
  - Research Site, Ponferrada
  - Research Site, Sabadell
  - Research Site, Salamanca
  - Research Site, Sant Boi de Llobregat
  - Research Site, Valencia
  - Research Site, Zaragoza
- Sweden (5):
  - Research Site, Helsingborg
  - Research Site, Karlskrona
  - Research Site, Lund
  - Research Site, Malmo
  - Research Site, Stockholm
- Taiwan (6):
  - Research Site, Kaohsiung City
  - Research Site, Keelung
  - Research Site, New Taipei City
  - Research Site, Taichung
  - Research Site, Taipei
  - Research Site, Taoyuan District
- United Kingdom (18):
  - Research Site, Belfast
  - Research Site, Birmingham
  - Research Site, Blackpool
  - Research Site, Bradford
  - Research Site, Chesterfield
  - Research Site, Corby
  - Research Site, Edinburgh
  - Research Site, Glasgow
  - Research Site, Kenilworth
  - Research Site, Liverpool
  - Research Site, London
  - Research Site, Middlesex
  - Research Site, Norwich
  - Research Site, Peterborough
  - Research Site, Romford
  - Research Site, Shipley
  - Research Site, Sidcup
  - Research Site, Wokingham

REFERENCES:
- [Derived] Muro S, Seki M, Hurst JR, Petullo D, Marshall J, Bowen K, Darken PF, Duncan EA, Megally A, Patel M. Triple Therapy with Budesonide/Glycopyrronium/Formoterol Fumarate Dihydrate versus Dual Therapies for Patients with COPD and Phenotypic Features of Asthma: A Pooled Post Hoc Analysis of KRONOS and ETHOS. Int J Chron Obstruct Pulmon Dis. 2024 Dec 12;19:2729-2737. doi: 10.2147/COPD.S478349. eCollection 2024. PMID 39691156
- [Derived] Singh D, Hurst JR, Martinez FJ, Rabe KF, Bafadhel M, Jenkins M, Salazar D, Dorinsky P, Darken P. Predictive modeling of COPD exacerbation rates using baseline risk factors. Ther Adv Respir Dis. 2022 Jan-Dec;16:17534666221107314. doi: 10.1177/17534666221107314. PMID 35815359
- [Derived] Rhodes K, Jenkins M, de Nigris E, Aurivillius M, Ouwens M. Relationship between risk, cumulative burden of exacerbations and mortality in patients with COPD: modelling analysis using data from the ETHOS study. BMC Med Res Methodol. 2022 May 25;22(1):150. doi: 10.1186/s12874-022-01616-7. PMID 35614467
- [Derived] Rabe KF, Martinez FJ, Ferguson GT, Wang C, Singh D, Wedzicha JA, Trivedi R, St Rose E, Ballal S, McLaren J, Darken P, Aurivillius M, Reisner C, Dorinsky P; ETHOS Investigators. Triple Inhaled Therapy at Two Glucocorticoid Doses in Moderate-to-Very-Severe COPD. N Engl J Med. 2020 Jul 2;383(1):35-48. doi: 10.1056/NEJMoa1916046. Epub 2020 Jun 24. PMID 32579807
- [Derived] Rabe KF, Martinez FJ, Ferguson GT, Wang C, Singh D, Wedzicha JA, Trivedi R, St Rose E, Ballal S, McLaren J, Darken P, Reisner C, Dorinsky P. A phase III study of triple therapy with budesonide/glycopyrrolate/formoterol fumarate metered dose inhaler 320/18/9.6 mug and 160/18/9.6 mug using co-suspension delivery technology in moderate-to-very severe COPD: The ETHOS study protocol. Respir Med. 2019 Oct-Nov;158:59-66. doi: 10.1016/j.rmed.2019.08.010. Epub 2019 Aug 22. PMID 31605923

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted in 26 countries between July 2015 and July 2019.
Pre-assignment Details: Subjects who successfully complete the Screening Period will then be randomized in a 1:1:1:1 scheme to BGF MDI 320/14.4/9.6 μg BID, BGF MDI 160/14.4/9.6 μg BID, BFF MDI 320/9.6 μg BID, or GFF MDI 14.4/9.6 μg BID, respectively.
Groups:
- BGF MDI 320/14.4/9.6 μg: Budesonide, Glycopyrronium, and Formoterol Fumarate Metered Dose Inhalation 320/14.4/9.6 μg
- BGF MDI 160/14.4/9.6 μg: Budesonide, Glycopyrronium, and Formoterol Fumarate Metered Dose Inhalation 160/14.4/9.6 μg
- GFF MDI 14.4/9.6 μg: Glycopyrronium, and Formoterol Fumarate Metered Dose Inhalation 14.4/9.6 μg
- BFF MDI 320/9.6 μg: Budesonide, Glycopyrronium, and Formoterol Fumarate Metered Dose Inhalation 320/9.6 μg
Period: Overall Study
Arm/Group | BGF MDI 320/14.4/9.6 μg | BGF MDI 160/14.4/9.6 μg | GFF MDI 14.4/9.6 μg | BFF MDI 320/9.6 μg
Started | 2157 | 2137 | 2143 | 2151
Completed | 1708 | 1713 | 1580 | 1643
Not Completed | 449 | 424 | 563 | 508
Not completed — Adverse Event | 118 | 113 | 147 | 138
Not completed — Lack of Efficacy | 103 | 102 | 171 | 135
Not completed — Withdrawal by Subject | 104 | 94 | 123 | 130
Not completed — Physician Decision | 23 | 33 | 38 | 28
Not completed — Major Protocol Deviation | 24 | 26 | 22 | 25
Not completed — Lost to Follow-up | 25 | 21 | 19 | 15
Not completed — Protocol Specified Criteria | 20 | 10 | 9 | 12
Not completed — Administrative Reasons | 12 | 9 | 11 | 5
Not completed — Randomized but not treated | 1 | 5 | 4 | 5
Not completed — enrolled in >1 studies | 18 | 11 | 19 | 15
Not completed — missing PI Signature | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: mITT population
Groups:
- Total: Total of all reporting groups
Arm/Group | BGF MDI 320/14.4/9.6 μg | BGF MDI 160/14.4/9.6 μg | GFF MDI 14.4/9.6 μg | BFF MDI 320/9.6 μg | Total
Number analyzed (Participants) | 2137 | 2121 | 2120 | 2131 | 8509
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.6 (7.6) | 64.6 (7.6) | 64.8 (7.6) | 64.6 (7.6) | 64.7 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 877 | 823 | 876 | 852 | 3428
  Male | 1260 | 1298 | 1244 | 1279 | 5081
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 400 | 393 | 426 | 401 | 1620
  Not Hispanic or Latino | 1690 | 1680 | 1649 | 1683 | 6702
  Unknown or Not Reported | 47 | 48 | 45 | 47 | 187
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 33 | 40 | 30 | 39 | 142
  Asian | 162 | 166 | 157 | 166 | 651
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 0 | 0 | 2
  Black or African American | 78 | 88 | 75 | 64 | 305
  White | 1819 | 1783 | 1808 | 1816 | 7226
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 43 | 44 | 50 | 46 | 183

OUTCOME MEASURES:

1. Primary Outcome: Adjusted Rate of Moderate or Severe Exacerbations
Description: Adjusted Rate of Moderate or Severe Exacerbations
Time Frame: 52-week treatment period
Population: mITT Population
Measure: Least Squares Mean (Standard Error); unit: Moderate or Severe Exacerbations
Arm/Group | BGF MDI 320/14.4/9.6 μg | BGF MDI 160/14.4/9.6 μg | GFF MDI 14.4/9.6 μg | BFF MDI 320/9.6 μg
Number analyzed (Participants) | 2137 | 2121 | 2120 | 2131
Moderate or Severe Exacerbations | 1.08 (0.04) | 1.07 (0.04) | 1.42 (0.05) | 1.24 (0.04)
Statistical Analysis 1: Comparison: BGF MDI 320/14.4/9.6 μg vs GFF MDI 14.4/9.6 μg; Test type: Superiority; p < 0.0001, Negative Binomial Regression; Rate Ratio = 0.76, 95% CI 2-sided [0.69 to 0.83]
Statistical Analysis 2: Comparison: BGF MDI 320/14.4/9.6 μg vs BFF MDI 320/9.6 μg; Test type: Superiority; p = 0.0027, Negative Binomial Regression; Rate Ratio = 0.87, 95% CI 2-sided [0.79 to 0.95]
Statistical Analysis 3: Comparison: BGF MDI 160/14.4/9.6 μg vs GFF MDI 14.4/9.6 μg; Test type: Superiority; p < 0.0001, Negative Binomial Regression; Rate Ratio = 0.75, 95% CI 2-sided [0.69 to 0.83]
Statistical Analysis 4: Comparison: BGF MDI 160/14.4/9.6 μg vs BFF MDI 320/9.6 μg; Test type: Superiority; p = 0.0020, Negative Binomial Regression; Rate Ratio = 0.86, 95% CI 2-sided [0.79 to 0.95]

2. Secondary Outcome: Time to First Moderate or Severe COPD Exacerbation
Description: Time to first moderate or severe COPD exacerbation (proportion with event reported as median time was not reached, statistical analyses are based upon time to event)
Time Frame: 52 Weeks
Population: mITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | BGF MDI 320/14.4/9.6 μg | BGF MDI 160/14.4/9.6 μg | GFF MDI 14.4/9.6 μg | BFF MDI 320/9.6 μg
Number analyzed (Participants) | 2137 | 2121 | 2120 | 2131
Participants | 1026 | 1013 | 1056 | 1085
Statistical Analysis 1: Comparison: BGF MDI 320/14.4/9.6 μg vs GFF MDI 14.4/9.6 μg; Test type: Superiority; p = 0.0035, Regression, Cox; Hazard Ratio (HR) = 0.880, 95% CI 2-sided [0.807 to 0.959]
Statistical Analysis 2: Comparison: BGF MDI 320/14.4/9.6 μg vs BFF MDI 320/9.6 μg; Test type: Superiority; p = 0.057, Regression, Cox; Hazard Ratio (HR) = 0.887, 95% CI 2-sided [0.814 to 0.966]
Statistical Analysis 3: Comparison: BGF MDI 160/14.4/9.6 μg vs GFF MDI 14.4/9.6 μg; Test type: Superiority; p = 0.0011, Regression, Cox; Hazard Ratio (HR) = 0.866, 95% CI 2-sided [0.794 to 0.944]
Statistical Analysis 4: Comparison: BGF MDI 160/14.4/9.6 μg vs BFF MDI 320/9.6 μg; Test type: Superiority; p = 0.0019, Regression, Cox; Hazard Ratio (HR) = 0.873, 95% CI 2-sided [0.801 to 0.951]

3. Secondary Outcome: Change From Baseline in Average Daily Rescue Ventolin HFA Use Over 24 Weeks
Description: Change from baseline in average daily rescue Ventolin HFA use over 24 weeks
Time Frame: 24 Weeks
Population: mITT Population
Measure: Least Squares Mean (95% Confidence Interval); unit: Puffs
Arm/Group | BGF MDI 320/14.4/9.6 μg | BGF MDI 160/14.4/9.6 μg | GFF MDI 14.4/9.6 μg | BFF MDI 320/9.6 μg
Number analyzed (Participants) | 1425 | 1389 | 1387 | 1426
Puffs | -1.2 [-1.3 to -1.1] | -1.0 [-1.2 to -0.9] | -0.7 [-0.8 to -0.5] | -0.8 [-0.9 to -0.7]
Statistical Analysis 1: Comparison: BGF MDI 320/14.4/9.6 μg vs GFF MDI 14.4/9.6 μg; Test type: Superiority; p < 0.0001, Linear Repeated Measures; Mean Difference (Final Values) = -0.51, 95% CI 2-sided [-0.68 to -0.34]
Statistical Analysis 2: Comparison: BGF MDI 320/14.4/9.6 μg vs BFF MDI 320/9.6 μg; Test type: Superiority; p < 0.0001, Linear Repeated Measures; Mean Difference (Final Values) = -0.37, 95% CI 2-sided [-0.54 to -0.20]
Statistical Analysis 3: Comparison: BGF MDI 160/14.4/9.6 μg vs GFF MDI 14.4/9.6 μg; Test type: Superiority; p < 0.0001, Linear Repeated Measures; Mean Difference (Final Values) = -0.35, 95% CI 2-sided [-0.53 to -0.18]
Statistical Analysis 4: Comparison: BGF MDI 160/14.4/9.6 μg vs BFF MDI 320/9.6 μg; Test type: Superiority; p = 0.0127, Linear Repeated Measures; Mean Difference (Final Values) = -0.22, 95% CI 2-sided [-0.39 to -0.05]

4. Secondary Outcome: Percentage of Subjects Achieving a MCID of 4 Units or More in SGRQ Total Score
Description: Percentage of subjects achieving a minimal clinically important difference (MCID) of 4 units or more in SGRQ (St. George's Respiratory Questionnaire) total score at Week 24
Time Frame: at Week 24
Population: mITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | BGF MDI 320/14.4/9.6 μg | BGF MDI 160/14.4/9.6 μg | GFF MDI 14.4/9.6 μg | BFF MDI 320/9.6 μg
Number analyzed (Participants) | 2119 | 2102 | 2096 | 2122
Participants | 1068 | 1024 | 893 | 949
Statistical Analysis 1: Comparison: BGF MDI 320/14.4/9.6 μg vs GFF MDI 14.4/9.6 μg; Test type: Superiority; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 1.358, 95% CI 2-sided [1.199 to 1.539]
Statistical Analysis 2: Comparison: BGF MDI 320/14.4/9.6 μg vs BFF MDI 320/9.6 μg; Test type: Superiority; p = 0.0005, Regression, Logistic; Odds Ratio (OR) = 1.246, 95% CI 2-sided [1.100 to 1.410]
Statistical Analysis 3: Comparison: BGF MDI 160/14.4/9.6 μg vs GFF MDI 14.4/9.6 μg; Test type: Superiority; p < 0.0004, Regression, Logistic; Odds Ratio (OR) = 1.283, 95% CI 2-sided [1.133 to 1.454]
Statistical Analysis 4: Comparison: BGF MDI 160/14.4/9.6 μg vs BFF MDI 320/9.6 μg; Test type: Superiority; p = 0.0103, Regression, Logistic; Odds Ratio (OR) = 1.177, 95% CI 2-sided [1.039 to 1.333]

5. Secondary Outcome: Time to Death (All Cause)
Description: Subject Deaths (all cause)
Time Frame: 52 Weeks
Population: ITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | BGF MDI 320/14.4/9.6 μg | BGF MDI 160/14.4/9.6 μg | GFF MDI 14.4/9.6 μg | BFF MDI 320/9.6 μg
Number analyzed (Participants) | 2137 | 2121 | 2120 | 2131
Participants | 28 | 39 | 49 | 34
Statistical Analysis 1: Comparison: BGF MDI 320/14.4/9.6 μg vs GFF MDI 14.4/9.6 μg; Test type: Superiority; p = 0.0111, Regression, Cox; Hazard Ratio (HR) = 0.544, 95% CI 2-sided [0.340 to 0.870]
Statistical Analysis 2: Comparison: BGF MDI 320/14.4/9.6 μg vs BFF MDI 320/9.6 μg; Test type: Superiority; p = 0.3401, Regression, Cox; Hazard Ratio (HR) = 0.782, 95% CI 2-sided [0.472 to 1.296]
Statistical Analysis 3: Comparison: BGF MDI 160/14.4/9.6 μg vs GFF MDI 14.4/9.6 μg; Test type: Superiority; p = 0.2690, Regression, Cox; Hazard Ratio (HR) = 0.789, 95% CI 2-sided [0.518 to 1.201]
Statistical Analysis 4: Comparison: BGF MDI 160/14.4/9.6 μg vs BFF MDI 320/9.6 μg; Test type: Superiority; p = 0.5918, Regression, Cox; Hazard Ratio (HR) = 1.134, 95% CI 2-sided [0.716 to 1.796]

6. Secondary Outcome: Rate of Severe COPD Exacerbations
Description: Rate of severe COPD exacerbations
Time Frame: 52 Weeks
Population: mITT Population
Measure: Least Squares Mean (Standard Error); unit: Severe Exacerbations
Arm/Group | BGF MDI 320/14.4/9.6 μg | BGF MDI 160/14.4/9.6 μg | GFF MDI 14.4/9.6 μg | BFF MDI 320/9.6 μg
Number analyzed (Participants) | 2137 | 2121 | 2120 | 2131
Severe Exacerbations | 0.13 (0.01) | 0.14 (0.01) | 0.15 (0.01) | 0.16 (0.01)
Statistical Analysis 1: Comparison: BGF MDI 320/14.4/9.6 μg vs GFF MDI 14.4/9.6 μg; Test type: Superiority; p = 0.6552, Negative Binomial Regression; Rate Ratio = 0.84, 95% CI 2-sided [0.69 to 1.03]
Statistical Analysis 2: Comparison: BGF MDI 320/14.4/9.6 μg vs BFF MDI 320/9.6 μg; Test type: Superiority; p = 0.0221, Negative Binomial Regression; Rate Ratio = 0.80, 95% CI 2-sided [0.66 to 0.97]
Statistical Analysis 3: Comparison: BGF MDI 160/14.4/9.6 μg vs GFF MDI 14.4/9.6 μg; Test type: Superiority; p = 0.2157, Negative Binomial Regression; Rate Ratio = 0.88, 95% CI 2-sided [0.72 to 1.08]
Statistical Analysis 4: Comparison: BGF MDI 160/14.4/9.6 μg vs BFF MDI 320/9.6 μg; Test type: Superiority; p = 0.0647, Negative Binomial Regression; Rate Ratio = 0.83, 95% CI 2-sided [0.69 to 1.01]

ADVERSE EVENTS:
Time Frame: Serious Adverse events were collected from the time subject signed Informed Consent to the time of the final follow-up telephone call. Adverse Events were collected from the time subject was randomized
Description: The Safety Population was defined as all subjects who were randomized to treatment and received at least 1 dose of the study drug
Arm/Group | BGF MDI 320/14.4/9.6 μg | BGF MDI 160/14.4/9.6 μg | GFF MDI 14.4/9.6 μg | BFF MDI 320/9.6 μg
All-Cause Mortality (participants affected / at risk) | 27/2144 | 42/2124 | 47/2125 | 35/2136
Serious Adverse Events (participants affected / at risk) | 426/2144 | 445/2124 | 433/2125 | 440/2136
Other Adverse Events (participants affected / at risk) | 337/2144 | 361/2124 | 292/2125 | 336/2136
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BGF MDI 320/14.4/9.6 μg (N=2144) | BGF MDI 160/14.4/9.6 μg (N=2124) | GFF MDI 14.4/9.6 μg (N=2125) | BFF MDI 320/9.6 μg (N=2136)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 202 (255) | 221 (263) | 219 (268) | 241 (299)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 14 (16) | 20 (20) | 20 (20) | 7 (7)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 9 (9) | 5 (5) | 9 (9)
Pulmonary emboism (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (3) | 5 (5) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 3 (3) | 4 (6)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 4 (4) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2) | 1 (1) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 0 (0) | 1 (1)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 0 (0) | 1 (1)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Laryngeal polyp (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Vocal cord leukoplakia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Bronchial secretion retention (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cystic lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasal turbinate hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pleurtitic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary calcification (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 61 (63) | 59 (64) | 35 (37) | 55 (57)
Sepsis (Infections and infestations) | 7 (8) | 5 (5) | 5 (5) | 3 (3)
Cellulitis (Infections and infestations) | 4 (4) | 6 (6) | 4 (4) | 3 (3)
Influenza (Infections and infestations) | 4 (4) | 2 (2) | 2 (2) | 7 (7)
Diverticulitis (Infections and infestations) | 3 (4) | 3 (3) | 3 (3) | 4 (5)
Bronchitis (Infections and infestations) | 2 (2) | 3 (3) | 4 (4) | 3 (3)
Urinary tract infection (Infections and infestations) | 1 (1) | 4 (4) | 2 (2) | 0 (0)
Respiratory tract infection (Infections and infestations) | 2 (3) | 2 (2) | 0 (0) | 2 (2)
Lung infection (Infections and infestations) | 1 (1) | 2 (2) | 1 (1) | 2 (2)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2) | 2 (2) | 1 (1)
Appendicitis (Infections and infestations) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Septic shock (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Erysipelas (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Pneumonia viral (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Staphylococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Anal abscess (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Peritonitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pneumonia pneumococcal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pulmonary tuberculosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Arthritis bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bacterial pyelonephritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchitis viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchopulmonary aspergillosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchopulmonary aspergillosis allergic (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bursitis infective (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Campylobacter infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Catheter site cellulitits (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cellulitis of male external genital organ (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis infective (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Colonic abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Emphysematous cholecystitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Encephalitis brain stem (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Endocarditis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Epididymitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis norovirus (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis salmonella (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis shigella (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
H1N1 influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Histoplasmosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infected bite (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infected dermal cyst (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infective exacerbation of bronshiectasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Laryngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Localised infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mastitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mastoiditis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Metapneumovirus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Micrococcus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oesophageal candidiasis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Osteomyelitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Otosalpingitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Perichondritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Periorbital cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia pseudomonal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Post procedural sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Soft tissue infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tracheobronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vaginal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 7 (8) | 10 (10) | 17 (18) | 7 (7)
Atrial fibrilation (Cardiac disorders) | 9 (9) | 8 (8) | 14 (15) | 3 (3)
Myocardial infarction (Cardiac disorders) | 5 (5) | 5 (5) | 7 (7) | 4 (4)
Coronary artery disease (Cardiac disorders) | 5 (5) | 5 (5) | 7 (7) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 5 (6) | 3 (3) | 5 (6) | 2 (2)
Cardiac arrest (Cardiac disorders) | 3 (3) | 1 (1) | 8 (8) | 0 (0)
Angina pectoris (Cardiac disorders) | 3 (3) | 0 (0) | 3 (3) | 5 (5)
Cardiac failure (Cardiac disorders) | 1 (1) | 3 (3) | 2 (2) | 3 (3)
Angina unstable (Cardiac disorders) | 3 (3) | 1 (1) | 3 (3) | 1 (1)
Cardiac failure acute (Cardiac disorders) | 1 (1) | 1 (1) | 4 (4) | 1 (1)
Cardiorespiratory arrest (Cardiac disorders) | 0 (0) | 1 (1) | 4 (4) | 2 (2)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 3 (3) | 1 (1) | 1 (1)
Stress cardiomyopathy (Cardiac disorders) | 0 (0) | 3 (3) | 1 (1) | 1 (1)
Arteriosclerosis coronary artery (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Atrial flutter (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Supraventricular tachycardia (Cardiac disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Arrhythmia (Cardiac disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Acute left ventricular failure (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Coronary artery occulsion (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pulseless electrical activity (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Ventricular fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Atriventricular block second degree (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac disorder (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardio-respiratory distress (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure chronic (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiogenic shock (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiovascular disorder (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiovascular insufficency (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Coronary artery stenosis (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertensive heart disease (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ischaemic cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Left ventricular failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mitral valve incompetence (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myocarditis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Right ventricular failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinus node dysfunction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tricuspid valve incompetence (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Trifascicular black (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 5 (5) | 2 (2) | 4 (4)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 1 (1) | 2 (2) | 3 (3)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 4 (4) | 1 (12)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1) | 0 (0) | 2 (2)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2) | 0 (0) | 1 (1)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Small cell lung caner (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Benign lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Malignant palate neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Oesophageal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Abdominal wall neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Adenosquamous cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Breast cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Breast cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Colon neopplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrooesophageal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hepatic cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Invasive breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Laryngeal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Metasteses to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Metastases to nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Metastatic bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oesophageal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Papillary renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Recosigmoid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tonsil cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 4 (4) | 3 (3) | 1 (1) | 5 (5)
Ankle fracture (Injury, poisoning and procedural complications) | 3 (3) | 0 (0) | 0 (0) | 3 (3)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 2 (2) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 2 (2) | 2 (2) | 0 (0) | 2 (2)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Abdominal wound dehiscene (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Multiple injuries (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Post procedural hemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Ulna fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Epicondylitis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Foreign body aspiration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Foreign body in gastrointestinal tract (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hand Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Humerous fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Jaw fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Limb traumatic amputation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Multiple fractures (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ocular procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Procedural pneumothorax (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pubis fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Radiation proctitis (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sternal fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Subdural hematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tendon rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Venomous bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wound decomposition (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 8 (8) | 2 (3) | 4 (4) | 3 (3)
Syncope (Nervous system disorders) | 2 (2) | 3 (3) | 1 (1) | 4 (4)
Cerebral infarction (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 5 (5)
Carotid artery stenosis (Nervous system disorders) | 2 (2) | 2 (2) | 0 (0) | 2 (2)
Siezure (Nervous system disorders) | 1 (1) | 4 (4) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Cerebellar infarction (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Ataxia (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Intracranial aneurysm (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Aphasia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Brain injury (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Carpal tunnel syndrome (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebrospinal fluid leakage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cervical radiculopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colloid brain cyst (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Embolic Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Guillain-Barre syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemorrhage intercranial (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hemorrhagic stroke (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hemiparesis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyopercapnic coma (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intercostal neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lacunar infarction (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Loss of consciousness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lumbar radiculopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Monparesis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myelopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ruptured cerebral aneurysm (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spinal claudication (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vocal cord paralysis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (3) | 2 (2) | 1 (1) | 2 (2)
Small intestine obstruction (Gastrointestinal disorders) | 2 (2) | 1 (1) | 2 (2) | 2 (2)
Abdonimal pain (Gastrointestinal disorders) | 1 (1) | 2 (2) | 2 (2) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Abdominal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Colitis ulcerative (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Diverticular perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Duodenal ulcenrn (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Anal fissure (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Colitis microscopic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diaphragmatic hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diverticulum (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Duodenal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastric ulcer perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemoroidal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemorrhoids thrombosed (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Impaired gastric emptying (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intestinal Infarction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Intestinal polyp (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mesenteric artery stenosis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Obstructive pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pharyngo-oesophageal diverticulum (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Varices oesophageal (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Death (General disorders) | 1 (1) | 4 (4) | 7 (7) | 2 (2)
Chest pain (General disorders) | 3 (3) | 4 (4) | 2 (2) | 2 (2)
Multiple organ dysfunction syndrome (General disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Sudden death (General disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 4 (4) | 1 (1) | 2 (2) | 4 (4)
Drug withdrawal syndrome (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Asthenia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Capsular contracture associated with breast implant (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Soft tissue inflamation (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sudden cardiac death (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Systemic inflammatory response syndrome (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 2 (2) | 3 (3) | 2 (2)
Peripheral arterial occlusive disease (Vascular disorders) | 3 (3) | 3 (3) | 0 (0) | 2 (2)
Deep vein thrombosis (Vascular disorders) | 4 (4) | 0 (0) | 0 (0) | 1 (1)
Hypertensive crisis (Vascular disorders) | 1 (1) | 2 (2) | 0 (0) | 2 (2)
Aortic aneurysm (Vascular disorders) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Aortic dissection (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Arteriosclerosis (Vascular disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Circulatory collapse (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypertensive urgency (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Iliac artery occlusion (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Peripheral Ischaemia (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Peripheral vascular disorder (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Accelerated hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aortic arteriosclerosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aortic stenosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peripheral artery occlusion (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral artery stenosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Shock Haemorrhagic (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Subclavian artery stenosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thrombophlebitis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Osteorthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 3 (3) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 2 (2) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Spinal ligament (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Synovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 2 (2) | 2 (2) | 3 (3) | 3 (3)
Cholelithiasis (Hepatobiliary disorders) | 3 (3) | 0 (0) | 4 (4) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Hepatic cirrohsis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Bile duct obstruction (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis Chronic (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatitis toxic (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 2 (2) | 1 (1) | 3 (3) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Renal colic (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Anuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemorrhage urinary tract (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lower urinary tract symptoms (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary bladder haemorrhage (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fluid overload (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Abnormal loss of weight (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diabetes melitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diabetes melitus inadequate control (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperlipidemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Impaired fasting glucose (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Obesity (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 0 (0) | 2 (2)
Iron deficiancy anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Anaemia macrocytic (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Immune thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alcohol withdrawal syndrome (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Schizoaffective disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Suicicide attempt (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Affective disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alcoholism (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hallucination (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Persistent depressive disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Retinal detachment (Eye disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Eyelid ptosis (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Retinal vascular thrombosis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Visual impairment (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Troponin increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Blood folate decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood magnesium decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Electrocradiogram ST-T change (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Electrocardiogram abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oxygen saturation decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Prothrombin time abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Allergy to arthropod sting (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Type I hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Endometrial hyperplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ovarian Cyst (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Scrotal cyst (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vaginal leukoplakia (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Swelling face (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Adrenal mass (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Goitre (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia streptococcal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cor pulmonale (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Non-Hodgkins lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Contussion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Penetrating abdominal trauma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumoconiosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wound evisceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Generalised tonic-clonic seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Erosive oesophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Large intestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Glomerulonephritis chronic (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 2 (2)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Retinal degeneration (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pnuemonia aspiration (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BGF MDI 320/14.4/9.6 μg (N=2144) | BGF MDI 160/14.4/9.6 μg (N=2124) | GFF MDI 14.4/9.6 μg (N=2125) | BFF MDI 320/9.6 μg (N=2136)
Nasopharyngitis (Infections and infestations) | 227 (290) | 239 (315) | 199 (255) | 234 (331)
Upper respiratory tract infection (Infections and infestations) | 123 (149) | 137 (176) | 102 (129) | 115 (154)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Drafts of any and all publications or presentations of this study must be submitted at least 30 days prior to submission for publication or presentation to Pearl Therapeutics for review, approval, and to ensure consistency. Pearl Therapeutics has the right to request appropriate modification to correct facts and to represent it's opinions, or the opinions of the publication committee, if these differ with the proposed publication.

DOCUMENTS (2):
  • Study Protocol (2019-06-21): https://cdn.clinicaltrials.gov/large-docs/67/NCT02465567/Prot_000.pdf
  • Statistical Analysis Plan (2019-04-30): https://cdn.clinicaltrials.gov/large-docs/67/NCT02465567/SAP_001.pdf